CLINICAL TRIAL: NCT05979441
Title: A Phase 3, Single-Arm, Multicenter, Open-label Extension of Study ARGX-113-2007 to Investigate the Long-term Safety, Tolerability, and Efficacy of Efgartigimod PH20 SC in Participants Aged 18 Years and Older With Active Idiopathic Inflammatory Myopathy
Brief Title: A Study to Assess the Long-term Safety and Efficacy of a Subcutaneous Formulation of Efgartigimod in Adults With Active Idiopathic Inflammatory Myopathy
Acronym: ALKIVIA+
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2011; 2022-502851-79-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myositis; Active Idiopathic Inflammatory Myopathy; Dermatomyositis; Polymyositis; Immune-Mediated Necrotizing Myopathy; Antisynthetase Syndrome
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Antisynthetase syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod PH20 SC (Experimental): Participants receiving efgartigimod PH20 subcutaneously
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous injection of Efgartigimod PH20 given by vials or prefilled syringe (PFS)

SUMMARY:
The main purpose of this study is to measure the long-term safety and tolerability of efgartigimod PH20 SC in adult participants with Idiopathic Inflammatory Myopathy (IIM) who previously participated in ARGX-113-2007.

The study consists of a treatment period where participants will receive efgartigimod PH20 SC for up to 51 months. The treatment period will be followed by a treatment-free safety follow-up period of 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Has completed trial ARGX-113-2007
* Being capable of providing signed informed consent and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and women of childbearing potential must have a negative urine pregnancy test at baseline before receiving the study drug

Exclusion Criteria:

* Intention to have major surgery during the study period or any other medical condition that has arisen since enrollment in study ARGX-113-2007, that in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Known hypersensitivity reaction to the study drug or 1 of its excipients
* Development of any malignancy, either new or recurrent, other than basal cell carcinoma of the skin, regardless of relatedness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and AESIs over time | Up to 53 months
  AE : adverse event ; SAE : serious adverse event ; AESI : adverse event of special interest.

SECONDARY OUTCOMES:
C-GTI comprising the AIS over time | Up to 51 months
  The Composite Glucocorticoid Toxicity Index (C-GTI) serves as a primary instrument to capture toxicities likely caused by glucocorticoid exposure and enables monitoring of long-term tolerability of glucocorticoids during prolonged use. The Aggregate Improvement Score (AIS) is an analytical scores generated from the weighted C-GTI. The AIS can be used to assess whether a new therapy is effective in reducing glucocorticoid toxicity over time; higher AIS scores are associated with less toxicity.
C-GTI comprising the CWS over time | Up to 51 months
  The Composite Glucocorticoid Toxicity Index (C-GTI) serves as a primary instrument to capture toxicities likely caused by glucocorticoid exposure and enables monitoring of long-term tolerability of glucocorticoids during prolonged use. The Cumulative Worsening Score (CWS) is an analytical score generated from the weighted C-GTI. The CWS is designed to assess cumulative glucocorticoid toxicity; higher scores indicate increased steroid toxicity.
C-GTI comprising the GTI-MD over time | Up to 51 months
  The Composite Glucocorticoid Toxicity Index (C-GTI) serves as a primary instrument to capture toxicities likely caused by glucocorticoid exposure and enables monitoring of long-term tolerability of glucocorticoids during prolonged use. The Glucocorticoid Toxicity Index-Metabolic Domains (GTI-MD) is an abbreviated GTI version limited to the 4 metabolic domains. A GTI-MD score of 0 indicates a low likelihood of toxicity in the assessed metabolic domains.
Prednisone dose reduction (average monthly dose) over time | Up to 51 months
TIS over time | Up to 51 months
  The total improvement score (TIS) assesses minimal, moderate, and major clinical response, and it is assessed using the ACR/EULAR criteria. The total score varies between 0 and 100, with higher scores indicating greater improvement.
Proportion of TIS responders (minimal, moderate, major) over time | Up to 51 months
  The total improvement score (TIS) assesses minimal, moderate, and major clinical response, and it is assessed using the ACR/EULAR criteria. The total score varies between 0 and 100, with higher scores indicating greater improvement
Individual CSMs of the TIS over time | Up to 51 months
  The total improvement score (TIS) assesses minimal, moderate, and major clinical response, and it is assessed using the ACR/EULAR criteria. The ACR/EULAR criteria calculate TIS using the 6 core set measure (CSMs): MDGA, PGA, MMT8, HAQ-DI, muscle enzymes, and extramuscular global assessment (assessed by the MDAAT).
Percentage of participants with clinically inactive disease | Up to 51 months
  Clinically inactive disease is defined as no evidence of disease activity, based on an Physician Global Assessment of Disease Activity (MDGA) and Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (MDAAT) of 0 and normal creatine kinase (CK) values for at least 12 weeks (at week 28 and every 24 weeks thereafter).
Percentage of participants with remission during the study | Up to 51 months
  Remission is defined as a clinically inactive disease for at least 24 weeks
PGI-S over time | Up to 51 months
  The Patient Global Impression of Severity (PGI-S) asks participants to rate the severity of their disease symptoms over the past 7 days on a 4-point Likert scale, where scores range from "no symptoms" to "severe."
CGI-S over time | Up to 51 months
  The Clinical Global Impression of Severity (CGI-S) asks the physician to rate the severity of the participant's disease on a 4-point Likert scale, where scores range from "no activity" to "severe".
Physical Functioning subscale and Physical Component Summary scores of the SF-36v2 over time | Up to 51 months
  The 36-Item Short Form Survey version 2 (SF-36v2) is a 36-item scale constructed to survey health-related quality of life in 8 domains.
EQ-5D-5L utilities over time | Up to 51 months
  The EQ-5D-5L questionnaire is a standardized test recognized by many health authorities as a generic measure of health status for clinical and economic appraisal. The descriptive system comprises 5 dimensions, each having 5 levels ranging from "No problem" to "Extreme problem".
EQ-5D-5L VAS over time | Up to 51 months
  The EQ-5D-5L questionnaire is a standardized test recognized by many health authorities as a generic measure of health status for clinical and economic appraisal. A visual analog scale (VAS) is included in the EQ-5D-5L, where participants will mark their health status from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Percent change from baseline in total IgG levels in serum over time | Up to 53 months
Incidence of ADA against efgartigimod (serum levels) over time | Up to 53 months
  ADA : anti-drug antibodies.
Proportion of participants achieving sustained low disease activity while on IMP, over time | Up to 51 months
  Sustained low disease activity is defined as a CGI-S score of "mild" or "no activity" and a PGI-S score of "mild" or "no symptoms" for at least 12 weeks.
Proportion of participants with low disease activity over time, while on IMP | Up to 51 months
  Low disease activity is defined as a CGI-S score of "mild" or "no activity" and a PGI-S score of "mild" or "no symptoms"
Proportion of participants with low disease activity who continue dosing every 2 weeks at week 52 and every 24 weeks thereafter | Up to 51 months
  Low disease activity is defined as a CGI-S score of "mild" or "no activity" and a PGI-S score of "mild" or "no symptoms"
Proportion of participants who have marked worsening during the period of dosing every 2 weeks | Up to 51 months
  Marked worsening is defined as a CGI-S score of "moderate" or "severe" and a PGI-S score of "moderate" or "severe"
Duration of dosing every 2 weeks | Up to 51 months

CONTACTS AND LOCATIONS:
Locations (78):
- United States (16):
  - Neuromuscular Clinical and Research Center - Neurology, Phoenix, Arizona
  - Attune Health Research, Inc, Beverly Hills, California
  - UCI Health - ALS and Neuromuscular Center - Neurology, Orange, California
  - UCSF Health - ALS and Neurodegenerative Disease Center - Dermatology, San Francisco, California
  - Yale Cancer Center-Yale University School Of Medicine, New Haven, Connecticut
  - UF Health - Rheumatology Medical Specialties Medical Plaza, Gainesville, Florida
  - Mayo Clinic - Florida - Neurology, Jacksonville, Florida
  - Emory Healthcare - Emory Clinic - Rheumatology, Atlanta, Georgia
  - Northwestern Medicine - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwell Health Physician Partners Rheumatology, Great Neck, New York
  - University of North Carolina (UNC) School of Medicine, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Austin Neuromuscular Center (National Neuromuscular Research Institute, PLLC), Austin, Texas
  - Nerve And Muscle Center Of Texas, Houston, Texas
- Argentina (3):
  - Framingham Centro Medico, La Plata
  - Centro Dermatologico Schejtman, San Miguel
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Tirol Kliniken - A.o. Landeskrankenhaus Innsbruck - Neurology, Innsbruck, Austria
- Belgium (2):
  - AZ Sint-Lucas - Campus Sint-Lucas - Neurology, Ghent
  - Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven
- Bulgaria (2):
  - Medical Centre Artmed, Plovdiv
  - Multiprofile hospital for active treatment Kaspela EOOD, Plovdiv
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Sichuan Provincial Academy of Medical Sciences and Sichuan Provincial People's Hospital, Chengdu
- Cyprus Institute of Neurology and Genetics, Nicosia, Cyprus
- Revmatologicky Ustav, Prague, Czechia
- Copenhagen University Hospital-Rigshospitalet University Hospital, Copenhagen, Denmark
- Reference Center Neuro-Muscular Diseases - CHU Paris Group Hospitalier La Pitie Salpetriere-Charles Foix, Paris, France
- Georgia (4):
  - Aversi Clinic, Tbilisi
  - LLC MediClub Georgia, Tbilisi
  - New Hospitals, Tbilisi
  - The First Medical Center, Tbilisi
- Germany (6):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte (CCM) - Rheumatology, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitatsmedizin Mannheim GmbH, Mannheim
  - Universitaetsklinikum Tuebingen (UKT), Tübingen
  - Klinikum der Universitaet Ulm, Ulm
- Greece (2):
  - National and Kapodistrian University of Athens - Eginition Hospital, Athens
  - ATTIKON University General Hospital - Neurology, Athens
- University College Dublin (UCD) - St. Vincent's University Hospital (SVUH), Dublin, Ireland
- Italy (6):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele Hospital, Milan
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara - Rheumatology, Pisa
  - Ospedale Sant'Andrea Hospital, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli - Neurology, Roma
  - Azienda sanitaria universitaria Friuli Centrale - ASUFC, Udine
- Japan (4):
  - Juntendo University Hospital, Bunkyō City
  - The University of Tokyo Hospital, Bunkyō City
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya
  - Wakayama Medical University Hospital, Wakayama
- Santaros University Clinic, Vilnius, Lithuania
- Hospital Angeles Clinica Londres, Mexico City, Mexico
- Amsterdam UMC Research BV, Amsterdam, Netherlands
- Peru (3):
  - Clinica San Juan de Dios - sede Arequipa - Rheumatology, Arequipa
  - Instituto Peruano Del Hueso Y La Articulacion Sac-Privado-Lima,Centro De Investigacion Iphar, Lima
  - Investigaciones Clinicas S.A.C., Lima
- Poland (2):
  - USK-WAM Centralny Szpital Weteranow - Szpital Kniniczny ul. Zeromskiego 113 - Rheumatology, Lodz
  - Centrum Wsparcia Badan Klinicznych Pomorskiego Uniwersytetu Medycznego w Szczecinie (CWBK PUM) - Rheumatology, Szczecin
- Centro Hospitalar do Porto - Hospital Santo Antonio, Porto, Portugal
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Institute of Rheumatology, Belgrade
- Seoul National University Hospital, Seoul, South Korea
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia - Neurology, Valencia
- Karolinska Universitestssjukhus Solna, Solna, Sweden
- Chung Shan Medical University Hospital, Taichung, Taiwan
- Thailand (5):
  - King Chulalongkorn Memorial Hospital - Neurology, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi hospital, Bangkok
  - Siriraj Hospital, Mahidol University of Internal medicine, Bangkok
  - Faculty Of Medicine, Khon Kaen University, Khon Kaen
- United Kingdom (3):
  - Aintree University Hospital - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - The Royal Free Hospital, London
  - Northern Care Allicance NHS Foundation Trust - Salford Royal - Rheumatology, Salford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study website — https://myositis-study.com/